CLINICAL TRIAL: NCT06872905
Title: Real-World Data Collection of the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis When Used in Covered Endovascular Reconstruction of the Aortic Bifurcation (CERAB) to Treat Aortoiliac Occlusive Disease
Status: Recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VBX 24-03
Record Dates: First submitted 2025-02-24; First posted 2025-03-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Aortoiliac Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- GORE VIABAHN® VBX Balloon Expandable Endoprosthesis: Patient was implanted with the VBX Device in the aortic and common iliac positions during the CERAB procedure.
  Interventions: Device: GORE VIABAHN® VBX Balloon Expandable Endoprosthesis (VBX)

INTERVENTIONS:
Device: GORE VIABAHN® VBX Balloon Expandable Endoprosthesis (VBX) — Treatment of Target Lesions with the VBX Device in the aortic and common iliac positions during the CERAB procedure.

SUMMARY:
The study will assess the safety and effectiveness of the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis ("VBX Device" or also referred to as "VBX Stent Graft") in a post approval setting and evaluate the quality of the use in covered endovascular reconstruction of the aortic bifurcation (CERAB) to treat Aortoiliac Occlusive Disease (AIOD).

DETAILED DESCRIPTION:
A minimum of 158 adult subjects will be enrolled at up to a minimum of 20 sites in the U.S. and Europe. Data will be collected retrospectively and found within existing site files at Baseline, Treatment, Discharge, Pre-12-Month Follow-up, 12-Month Follow-Up, Subsequent Follow-Up Visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient treated with covered endovascular reconstruction of the aortic bifurcation (CERAB) procedure for aortoiliac occlusive disease (AIOD).
2. Patient was implanted with the VBX Device in the aortic position during a CERAB procedure.
3. Patient was treated with the CERAB procedure a minimum of 1 year before enrollment date.
4. Age ≥18 years at the time of CERAB procedure.
5. Obtain patient informed consent or waiver according to local Institutional Review Board (IRB)/Ethics Committee (EC) -

Exclusion Criteria:

1. Patient with prior stenting in the aortic or common iliac artery at the time of CERAB procedure.
2. Patient treated with concomitant chimney procedure at time of CERAB procedure (e.g., inferior mesenteric artery, renal artery).
3. Participation in another drug or device investigational study at the time of the CERAB procedure date that can confound the study endpoints.

   -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As described in the background section, patients with aortoiliac occlusive disease are treated with various surgical and endovascular therapies to improve arterial blood flow to the lower extremity. This study will retrospectively evaluate a population of patients that have had covered endovascular reconstruction of the aortic bifurcation (CERAB) with GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis.
  The study has been designed with standard eligibility criteria to evaluate the safety and effectiveness of the VBX Device when used in a CERAB for an aortoiliac occlusive disease patient population.
  Considering the nature of aortoiliac occlusive disease, elderly patients (≥ 65 years old) can represent a significant number of patients enrolled in this study. This population can include patients with cognitive disorder or severe dementia.
  According to EU regulation, elderly patients are considered vulnerable population. However, considering the retrospective nature of the study design, t
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-08-16 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: 1-Year Primary patency (hypothesis testing) | 1-Year
  Proportion of patients maintaining primary patency at 1 Year
Primary Safety Endpoint: 30-day Morbidity (hypothesis testing) | 30-Day
  Proportion of patients experiencing any major adverse cardiovascular event (i.e. myocardial infarction, cerebrovascular accident) or event requiring reintervention.

SECONDARY OUTCOMES:
Technical Success | At index procedure
  Proportion of patients with technical success
Mortality | 30-Day
  Proportion of patients with all cause death
Device Integrity | 1 year
  Proportion of patients achieving Primary Patency
Primary assisted patency | 1 year
  Proportion of patients achieving Primary Assisted patency
Secondary patency | 1 year
  Proportion of patients achieving Secondary Patency
Freedom from Target Lesion Revascularization | 1 year
  Proportion of patients achieving freedom from Target Lesion Revascularization
Survival | 1 Year
  Proportion of patients survival
Freedom from Clinically-Driven Target Lesion Revascularization | 1 year
  Proportion of patients achieving freedom from Clinically-Driven Target Revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Ann O'Banion, M.D., Principal Investigator — University of California, San Francisco; Michele Antonello, M.D., Principal Investigator — Azienda Ospedaliero-Universitaria di Padova
Locations (18):
- United States (12):
  - University of California, Fresno, California
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Rutgers, New Brunswick, New Jersey
  - Research Foundation SUNY Buffalo, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - The University of Texas Austin, Austin, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Marshfield Hospital, Marshfield, Wisconsin
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Padova, Padua
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (2):
  - Amsterdam UMC Research BV, Amsterdam
  - Franciscus, Rotterdam
- Hospital General Universitario de Alicante, Alicante, Spain
- Greater Glasgow Health Board, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No